CLINICAL TRIAL: NCT02038322
Title: The Stork™ Conception System (OTC) Clinical Trial: Semen Collection, Placement and Delivery
Brief Title: The Stork OTC: Collection, Placement & Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rinovum Women's Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ER-000025
Record Dates: First submitted 2013-10-28; First posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Safety and Usability
Keywords: OTC Home Use Conception Aid Cervical Cap Insemination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The Stork (No Intervention): Device - The Stork - complete kit (Conceptacle and Applicator)
  Interventions: Device: The Stork - Conception Aid

INTERVENTIONS:
Device: The Stork - Conception Aid
  Other Names: The Stork

SUMMARY:
This is a clinical study designed to validate the usability and safety of the over-the-counter (OTC) device by obtaining feedback in a home use environment regarding ease of use of The Stork™ Conception System and the instructions for use. In addition to usability, results for safety, including vaginal

DETAILED DESCRIPTION:
Female participants will undergo a baseline pelvic examination. Participating couples will be given The Stork™ Conception System (OTC), including Instructions for Use, the questionnaire and two ziplock bags. The device will be used in accordance with the instructions for use. Participants will use the Conceptacle as a collection condom during sexual intercourse. Participants will remove the Cervical Cap from the Sheath of the Conceptacle and discard the Sheath. Participants will then load the Cervical Cap into the Applicator for insertion, placement and deployment of the device. Participants will wash the applicator with soap and water and place it in the double zip lock bags. During the time the cervical cap is inserted, normal activity will be recommended with the exception of having intercourse. The female participants will leave the conception cap inserted for a period of time between 4 and 12 hours, return to the investigator's office for examination, remove the Cervical Cap, and undergo a follow up pelvic examination. Participants will be asked to complete the study and the questionnaire within 3 days of receiving the study packet. As a result, this study could take up to 4 days to complete per enrolled couple.

ELIGIBILITY:
Inclusion Criteria:

* Literacy must be in English (able to understand Informed Consent)
* In general good health
* Heterosexual, monogamous couples, of any race or ethnicity, who are sexually active (as a couple)
* 18 - 50 years of age
* REALM-SF Test Results demonstrate 6th grade literacy or above
* Past experience with using condoms
* Trying to conceive or using a non-vaginal birth control with which they do not normally use a condom.
* Signed Informed Consent

Exclusion Criteria:

* Vaginal prolapsed (female)
* Hysterectomy (female)
* Erectile Dysfunction (male)
* Colposcopy with biopsy surgery within the last three (3) months (female)
* Treatment for dysplasia surgery within the last three (3) months (female)
* Vaginal/cervical surgery within the last three (3) months (female)
* Current Pregnancy (female)
* Unable to read and understand English

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Efficacy -Primary endpoint part 1 - Collection | 1-3 days
  The primary endpoint of the study is comprised of 3 parts. It is binary, in the sense that if all of the three parts are "passed" then the endpoint is met for that couple. If any part of the endpoint is not met then the endpoint for that couple is not met. The three parts of the endpoint are:
  P1: Participants indicate ability to collect and contain semen using the Conceptacle™.
  The examinations will occur 4-12 hours after device insertion.
Efficacy - Primary endpoint part 2 - Placement | 4-12 hrs
  The primary endpoint of the study is comprised of 3 parts. It is binary, in the sense that if all of the three parts are "passed" then the endpoint is met for that couple. If any part of the endpoint is not met then the endpoint for that couple is not met.
  P2: Successful placement of the cervical cap as determined by physical examination.
Primary endpoint part 3 -Safety | 4-12 hrs
  The primary endpoint of the study is comprised of 3 parts. It is binary, in the sense that if all of the three parts are "passed" then the endpoint is met for that couple. If any part of the endpoint is not met then the endpoint for that couple is not met.
  P3: Participants use the device without any evidence of damage to the female participants' genital tract as depicted by physician examination.

SECONDARY OUTCOMES:
Secondary Endpoint | up to 3 days
  Secondary Objectives: Pass/Fail Answers to the specific questions Male 1-3 and Female 1-4 on the CRF will be compiled descriptively to indicate participant success during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Pelekanos, OB-GYN, Principal Investigator — Forbes Regional Hospital
Locations (1):
- Forbes Regional Hospital, Monroeville, Pennsylvania, United States